CLINICAL TRIAL: NCT02698943
Title: Evaluation of Glistenings and Posterior Capsule Opacification Following Envista MX60 Intraocular Lens Implantation
Brief Title: Glistenings and PCO Evaluation for the Envista MX60
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Other Study IDs: 320/2-3-2016
Record Dates: First submitted 2016-03-02; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Cataract
Keywords: cataract; intraocular lens; posterior capsule opacification; glistening; ENVISTA
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Participants who underwent phacoemulsification surgery and implantation of the Envista MX-60 IOL
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Phacoemulsification for cataract extraction with Envista MX-60 implantation

SUMMARY:
Posterior capsule opacification (PCO) and glistenings development is among the primary reasons for sub-optimal visual capacity following cataract extraction surgery. Primary objective of this study is to evaluate the incidence of PCO and glistenings of the popular envista MX-60 intraocular lens (Bausch + Lomb) in a random sample of cataract patients who underwent phacoemulsification at least 1 year prior to their enrollment at the study

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of senile cataract with stage 3 nuclear opalescence according to the Lens Opacities Classification System III (LOCS-3) grading scale

Exclusion Criteria:

Endothelial cell count less than 1900, glaucoma, IOP-lowering medications, former incisional surgery, former diagnosis of corneal disease, diabetes or autoimmune diseases

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with senile cataract
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Glistenings | 1 year
  Evaluation of glistenings using Scheimpflug analysis
Posterior capsule Opacification (PCO) | 1 year
  Evaluation of PCO using EPCO software

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Assistant Professor

IPD SHARING:
Plan to Share IPD: No